CLINICAL TRIAL: NCT07133685
Title: Evaluation of Serum IL-7 as a Biomarker in Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Emad Eldin Abd Allah Mahran, residant doctor at Assiut university hospital, Assiut University
Other Study IDs: Serum IL-7 Breast Cancer
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: Female patients diagnosed with Breast cancer based on pathological and radiological confirmation.

SUMMARY:
Breast cancer is one of the most commonly diagnosed cancers and leading cause of cancer-related mortality in women worldwide, posing a serious threat to their health (1).

It is a heterogeneous disease, characterized by varying molecular subtypes such as hormone receptor-positive (HR+), human epidermal growth factor receptor 2 (HER2-positive), and triple-negative breast cancer (TNBC) (2).

Breast cancer develops as a result of several internal and external factors (3-5). Poor lifestyle choices, environmental factors, and social-psychological factors are all linked to its occurrence. It has been demonstrated that 5% to 10% of breast cancers can be attributed to genetic mutations and family history, while 20% to 30% of breast cancers can be attributed to factors that may be modifiable (6). An early and accurate diagnosis is essential for effective treatment and improved patient survival.

The human immune system plays a fundamental role in the defense against malignant diseases by recognizing and eliminating cancerous cells at the early stages of tumor development. Many research has been conducted on various cytokines to assess their role in the development of various tumors.

IL-7 is an essential cytokine for the adaptive immune system, which is crucial for the development of B cells, the proliferation and survival of memory T cells and naive T cells, as well as the development of thymic T cells (7).

IL-7 action is realized through two main signaling pathways: (Jak-Stat and PI3K-Akt) (8). Through these pathways, it has an impact on the development, survival, proliferation, differentiation and maturity of immune cells such as T-lymphocytes, B-lymphocytes, and natural killer cells (9).

IL-7 has strong immunomodulatory act on tumor cells and exerts anti-tumor effects by enhancing tumor eradication or adoptive immunity (10).

However, IL-7 may also facilitate tumor progression by activating the same downstream AKT pathways .

ELIGIBILITY:
Inclusion Criteria:

* Female patients diagnosed with Breast cancer based on pathological and radiological confirmation.
* Age > 18

Exclusion Criteria:

* Male
* Patients diagnosed with other malignant diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female patients
Study Population: Female patients diagnosed with Breast cancer based on pathological and radiological confirmation.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
concentration of the serum level of IL-7 in patients with breast cancer | baseline
  concentration of the serum level of IL-7 in patients with breast cancer